CLINICAL TRIAL: NCT02106195
Title: A Phase 2a, Open-label Study to Evaluate the Safety and Tolerability of KD025 [Belumosudil] Treatment in Subjects With Moderately Severe Psoriasis Vulgaris Who Have Failed First-line Therapy
Brief Title: A Safety and Tolerability Study of Belumosudil (KD025) Treatment in Subjects With Moderately Severe Psoriasis Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kadmon Corporation, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD025-205
Record Dates: First submitted 2014-04-02; First posted 2014-04-08 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Psoriasis Vulgaris
MeSH Terms: interventions — belumosudil; KD025

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Belumosudil 200 mg (Experimental): Belumosudil 200 mg (two 100 mg capsules) orally once daily for 28 days
  Interventions: Drug: Belumosudil

INTERVENTIONS:
Drug: Belumosudil
  Other Names: Rezurock (brand name); KD025; SLx-2119

SUMMARY:
The primary objective is to assess the safety and tolerability of 200 mg of belumosudil administered orally once daily for 28 days.

DETAILED DESCRIPTION:
This will be a Phase 2a, open-label, single-arm, safety and tolerability study of belumosudil given daily for treatment of psoriasis.

Eight subjects with moderately severe psoriasis who have failed at least 1 line of systemic therapy will be enrolled.

Treatment Period Eligible subjects who have failed at least 1 line of systemic therapy will be entered and treated for 4 weeks (28 days) with 200 mg of belumosudil given orally once daily (QD).

Subjects will undergo medical history evaluations, physical examinations, vital sign measurements, weight, adverse event assessments, concomitant medication assessments, and laboratory testing including but not limited to blood sample collection for hematology and chemistry, urinalysis, coagulation, lipid panel, electrocardiogram, pregnancy test for females of childbearing potential, testing with the Psoriasis Area and Severity Index (PASI) scale and Physician Global Assessment (PGA) scale, and pharmacokinetic sampling.

Follow-up Period:

Visit will occur 4 weeks after the last dose of study drug in the Treatment Period of the study. This visit must be done within ± 3 days of the scheduled visit. The same assessments will be performed as in the Treatment Period.

The duration of the study is 12 weeks: up to 4 weeks for screening, 4 weeks of treatment, and 4 weeks of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of moderately severe plaque psoriasis that has been stable for 6 months and has failed at least one line of systemic therapy and is a candidate for additional systemic therapy.
* Had a PASI of ≥12
* At least 10% of body surface area that is affected by plaque psoriasis.
* Willing to avoid tanning devices or sun bathing.
* Willing to forgo systemic and topical treatments for psoriasis during the course of the study.
* Adequate bone marrow function
* Negative urine pregnancy test (for women of childbearing potential)
* Agree to use a highly effective method of birth control (< 1% per year failure rate) during the study and for 1 month after the termination of the study.
* Willing to complete all study measurements and assessments in compliance with the protocol.

Exclusion Criteria:

* Non-plaque or drug-induced psoriasis
* Currently using corticosteroid or immunosuppressive therapy except for Class 5 or weaker topical corticosteroids to the face, groin, or scalp
* Using any topical therapy except for the following:

  1. Class 5 or weaker steroids and phototherapy for 4 weeks prior to study entry
  2. Immunosuppressive therapies for 4 weeks prior to study entry
  3. Methotrexate, acitretin, or cyclosporine for 4 weeks prior to study entry
  4. Biologic therapies for 3 months prior to study entry.
* Concomitant condition requiring treatment with moderate to high dose steroids in the 12 weeks prior to screening.
* Viral, fungal, or bacterial skin infection.
* Pregnant or lactating woman.
* Currently participating in another study with an investigational drug or within 28 days of study entry
* History or other evidence of severe illness or any other conditions that would make the subject, in the opinion of the investigator, unsuitable for the study
* History or presence of any of the following:

  1. Hepatic disease and or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 1.5 × the upper limit of normal (ULN) at screening
  2. Renal disease and/or serum creatinine > 1.5xULN at screening
* Has QTc(f) intervals of > 450 msec at the screening or pre-dose ECG
* Subject is receiving any drugs known to prolong the QTc interval, including any anti-arrhythmic medications within 2 weeks prior to screening
* Subject is receiving any drug that is a strong CYP enzyme inhibitor
* Subject is receiving any concomitant systemic drug that is metabolized by CYP enzyme
* Previous exposure to KD025 or known allergy/sensitivity to KD025 or any other ROCK-2 inhibitor.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Irvine Health, Dept of Dermatology, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Open-label, Phase 2a, single-arm study of subjects with moderately severe plaque psoriasis who had been stable for 6 months and had failed at least 1 line of systemic therapy. Subjects were recruited at 1 site in the U.S.
Pre-assignment Details: Screening assessments occurred within 28 days prior to assignment and included informed consent, medical/demographic history, physical exam, vital signs, clinical laboratory tests, ECG, urine pregnancy, skin punch biopsy, PK, Psoriasis Area and Severity Index (PASI) scoring, Physician Global Assessment (PGA) scoring, and concomitant AE assessments.
Groups:
- Belumosudil 200 mg PO QD: 8 subjects with moderately severe psoriasis who had failed at least 1 line of systemic therapy administered belumosudil 200 mg orally QD for 4 weeks
Period: Overall Study
Arm/Group | Belumosudil 200 mg PO QD
Started | 8
Completed | 5 (Includes all 3 periods of study: Screening, Treatment, Post-treatment)
Not Completed | 3
Not completed — Adverse Event | 2
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Groups:
- Belumosudil 200 mg PO QD: Belumosudil 200 mg (two 100 mg capsules) orally once daily for 28 days
Arm/Group | Belumosudil 200 mg PO QD
Number analyzed (Participants) | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.6 (10.31)
Age, Customized [Median (Full Range); unit: years] | 49.5 [31 to 57]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index (kg/m^2)
  kg/m^2 | 29.42 (6.539)
BMI [Median (Full Range); unit: kg/m^2] — Body mass index (kg/m^2)
  kg/m^2 | 27.61 [21.2 to 41.0]

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Adverse Events as a Measure of Safety and Tolerability
Description: To evaluate the safety and tolerability of 200 mg of belumosudil administered PO QD to subjects for treatment of psoriasis
Time Frame: Up to 12 weeks:Up to 4 weeks screening (depending on signed informed consent + 4 weeks treatment + 4 weeks follow-up
Population: Safety Population: All subjects who received at least 1 dose of belumosudil 200 mg
Measure: Count of Participants; unit: Participants
Groups:
- Belumosudil 200 mg PO QD: Subjects who received at least 1 dose of belumosudil 200 mg orally daily
Arm/Group | Belumosudil 200 mg PO QD
Number analyzed (Participants) | 8
Participants
  All AEs | 4
  Related AEs | 1
  Grade ≥3 AEs | 1
  Grade ≥3 Related AEs | 0
  Grade 4 AEs | 0
  Deaths | 0
  SAEs | 1
  Related SAEs | 0
  AEs leading to discontinuation | 2

2. Secondary Outcome: Efficacy: Change in Overall PASI (Psoriasis Area and Severity Index) From Baseline to Week 4 and Week 8
Description: The Psoriasis Area and Severity Index (PASI) is a composite score based on the degree of effect on body surface area of psoriasis and the extension of erythema (reddening), induration (thickness), desquamation (scaling) of the lesions and area affected as observed on the day of examination. The severity of each sign was assessed using a 5-point scale, where 0=no symptoms, 1=slight, 2=moderate, 3=marked, 4=very marked. The PASI score ranges from 0 to 72, where 0 indicates no psoriasis and 72 indicates very severe psoriasis.
  The measures are the changes in PASI score at Week 4 from baseline and Week 8 from baseline. Negative changes are favorable; positive changes are unfavorable.
Time Frame: 8 weeks: 4-week (28-day) treatment + 4-week (28-day) follow-up
Population: All 8 subjects who received belumosudil 200 mg PO QD. 7 subjects available at follow-up visit.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Belumosudil 200 mg PO QD: Subjects receiving 200 mg of belumosudil daily
Arm/Group | Belumosudil 200 mg PO QD
Number analyzed (Participants) | 8
Score on a scale
  Baseline (Day 1) | 17.5 (8.41)
  Week 4 (Day 28) | 16.3 (9.49)
  Change from Baseline to Week 4 | -1.1 (3.04)
  Week 8 (Day 56): number analyzed (Participants) | 7
  Week 8 (Day 56) | 14.7 (3.41)
  Change from Baseline to Week 8: number analyzed (Participants) | 7
  Change from Baseline to Week 8 | 0.0 (1.54)
Statistical Analysis 1: Comparison: Belumosudil 200 mg PO QD; Test type: Superiority — Change from Baseline to Day 28; p = 0.324, t-test, 2 sided; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-3.7 to 1.4], Standard Deviation 3.04

3. Secondary Outcome: Efficacy: Physician Global Assessment (PGA) at Week 4 and Week 8
Description: PGA score after treatment with belumosudil 200 mg PO QD at 4 weeks (28 days treatment) and at 8 weeks (additional 4 weeks follow-up).
  Categories: 100% = clear; 75% to 99% clearing (Excellent) = marked improvement, nearly normal skin texture, some erythema may be present; 50% to 74% clear (Good) = moderate improvement, plaque has cleared to point of small scattered papules with normal intervening epidermis; 25% to 49% clearing (Fair) = slight improvement, decrease in scaling and softening of plaque; 0% to 24% clearing (Poor) = little or no change in scaling, erythema, or plaque elevation; Worse
Time Frame: 8 weeks: 4-week (28-day) treatment + 4-week (28-day) follow-up
Population: All 8 subjects had PGA scoring at Day 29 and at the follow-up visit (30 days after last dose of study drug)
Measure: Count of Participants; unit: Participants
Groups:
- Belumosudil 200 mg PO QD: Subjects receiving belumosudil 200 mg orally once daily for up to 28 days
Arm/Group | Belumosudil 200 mg PO QD
Number analyzed (Participants) | 8
Participants
  4 weeks: 75% to 100% | 0
  4 weeks: 50% to 74% clearing | 1
  4 weeks: 25% to 49% clearing | 1
  4 weeks: 0 to 24% clearing | 4
  4 weeks: Worse | 2
  8 weeks: 75% to 100% | 0
  8 weeks: 50% to 74% clearing | 0
  8 weeks: 25% to 49% clearing | 0
  8 weeks: 0% to 24% clearing | 6
  8 weeks: Worse | 1
  8 weeks: Missing (no data) | 1

4. Secondary Outcome: PK: Cmax and Cmin
Description: Pharmacokinetic measures:
  Cmax = maximum observed plasma concentration; Cmin = minimum observed plasma concentration over 1 dosing period; KD025 = Parent Drug KD025; M1 = Metabolite KD025 M1; KD025 M2 = Metabolite M2.
  Day 1 Cmax: 8 subjects each in KD025 and M2, and 6 subjects in M1. Day 28 Cmax: 4 subjects each in KD025 and M2, and 1 subject in M1.
  Day 1 Cmin: 8 subjects each in KD025 and M2, and 3 subjects in M1. Day 28 Cmin: 4 subjects each in KD025 and M2, and 1 subject in M1.
Time Frame: Measured at Baseline (Day 1) and Week 4 (28 days): predose (0), 1, 2, 4, 8, and 24 hours post-dose
Population: One subject excluded from all the descriptive statistics due to a mix-up of samples between predose and 4 hours (KD025, M1 and M2); Two subjects had no measurable concentrations observed in their profiles for M1 at Day 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Parent Drug KD025: Study drug belumosudil
- Metabolite M1: Metabolite KD025 M1 of parent drug KD025.
- Metabolite M2: Metabolite KD025 M2 of parent drug KD025.
Arm/Group | Parent Drug KD025 | Metabolite M1 | Metabolite M2
Number analyzed (Participants) | 8 | 6 | 8
ng/mL
  Cmax: Day 1 | 1240 (704) | 21.3 (10.9) | 221 (165)
  Cmax: Day 28: number analyzed (Participants) | 4 | 1 | 4
  Cmax: Day 28 | 810 (475) | 15.0 (NA) — Standard Deviation is not available since only 1 participant was analyzed for the assessment. | 131 (152)
  Cmin: Day 1: number analyzed (Participants) | 8 | 3 | 8
  Cmin: Day 1 | 59.6 (29.3) | 18.7 (9.16) | 21.1 (6.13)
  Cmin: Day 28: number analyzed (Participants) | 4 | 1 | 4
  Cmin: Day 28 | 35.9 (22.9) | 10.7 (NA) — Standard Deviation is not available since only 1 participant was analyzed for the assessment. | 17.6 (7.36)

5. Secondary Outcome: PK: AUC(0-24) and AUC(Inf)
Description: Pharmacokinetic measures:
  AUC(0-24) = area under concentration time-curve from pre-dose (time 0) to 24 hours post-dose; AUC(inf) = area under concentration time-curve extrapolated from Day 1 to infinity; KD025 = Parent Drug KD025; M1 = Metabolite KD025 M1; KD025 M2 = Metabolite M2.
Time Frame: Measured at Baseline (Day 1) and Week 4 (28 days): predose (0), 1, 2, 4, 8, and 24 hours post-dose
Population: AUC(0-24) Day 1: 7 subjects in KD025 and 3 subjects in M2. AUC(0-24) Day 28: 4 subjects in KD025 and 2 subjects in M2. AUC(inf): 6 subjects in KD025 and 3 subject in M2. Neither AUC(0-24) nor AUC(inf) were calculated for M1.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Parent Drug KD025 | Metabolite M2
Number analyzed (Participants) | 7 | 7
ng*hr/mL
  AUC(0-24): Day 1: number analyzed (Participants) | 7 | 3
  AUC(0-24): Day 1 | 7360 (3180) | 1040 (545)
  AUC(0-24): Day 28: number analyzed (Participants) | 4 | 2
  AUC(0-24): Day 28 | 5500 (3790) | 162 (2320)
  AUC(inf) from Day 1: number analyzed (Participants) | 6 | 3
  AUC(inf) from Day 1 | 8230 (3600) | 1120 (680)

6. Secondary Outcome: PK: Tmax
Description: Pharmacokinetic measure:
  Tmax = time of maximum observed plasma concentration. Day 1 Tmax: 7 subjects each in KD025 and M2, and 5 subjects in M1. Day 28 Tmax: 4 subjects each in KD025 and M2, and 1 subject in M1.
Time Frame: Measured at Baseline (Day 1) and Week 4 (28 days): predose (0), 1, 2, 4, 8, and 24 hours post-dose
Population: Day 1: 7 subjects each in KD025 and M2, and 5 subjects in M1. Day 28: 4 subjects each in KD025 and M2, and 1 subject in M1.
Measure: Median (Full Range); unit: hours
Arm/Group | Parent Drug KD025 | Metabolite M1 | Metabolite M2
Number analyzed (Participants) | 7 | 5 | 7
hours
  Tmax: Day 1 | 2.00 [1.00 to 7.92] | 2.00 [1.00 to 2.00] | 2.00 [1.00 to 7.92]
  Tmax: Day 28: number analyzed (Participants) | 4 | 1 | 4
  Tmax: Day 28 | 4.00 [1.00 to 4.13] | 4.00 [4.00 to 4.00] | 4.00 [1.00 to 4.13]

7. Secondary Outcome: PK: t(1/2)
Description: KD025 = Parent Drug KD025; KD025 M2 = Metabolite M2; t(1/2) = apparent terminal elimination half-life
Time Frame: Measured at Baseline (Day 1) and Week 4 (28 days): predose (0), 1, 2, 4, 8, and 24 hours post-dose
Population: One subject was excluded from all descriptive statistics due to a mix-up of samples between pre-dose and 4 hours on Day 1.
  Three subjects were excluded from day 28 statistics due to varying protocol deviations. Four additional subjects were excluded from M1 Day 28. No data were collected for Metabolite M1.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Parent Drug KD025 | Metabolite M2
Number analyzed (Participants) | 6 | 3
hours
  t(1/2): Day 1 | 6.08 (0.681) | 4.25 (3.95)
  t(1/2): Day 28: number analyzed (Participants) | 3 | 1
  t(1/2): Day 28 | 5.27 (0.692) | 2.26 (NA) — Standard Deviation not available since only 1 participant was analyzed for the assessment.

ADVERSE EVENTS:
Time Frame: 12 weeks: up to 4 weeks for screening, 4 weeks of treatment, and 4 weeks of follow-up.
Description: The National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 4.03 was used. The Clinical Symptom and Adverse Event Grading scale was used for grading toxicities.
Groups:
- Belumosudil 200 mg PO QD: Subjects who received belumosudil 200 mg orally daily
Arm/Group | Belumosudil 200 mg PO QD
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 1/8
Other Adverse Events (participants affected / at risk) | 4/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil 200 mg PO QD (N=8)
Nausea (Gastrointestinal disorders) | 1 (1) — Same subject had SAE
Vomiting (Gastrointestinal disorders) | 1 (2) — Same subject had SAE
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 (1) — Same subject had SAE
Nephrolithiasis (Renal and urinary disorders) | 1 (1) — Same subject had SAE
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Belumosudil 200 mg PO QD (N=8)
Transaminase increased (Investigations) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (2)
Anastomotic ulder (Injury, poisoning and procedural complications) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Tooth ache (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results. The sponsor cannot require changes to the study results in the communication except to remove sponsor's confidential information. Sponsor cannot unilaterally extend the embargo.